CLINICAL TRIAL: NCT03061162
Title: Phase II Study of Pulsed Low Dose Rate Radiation Therapy for Gastric Cancer Patients With Peritoneal Metastasis
Brief Title: Pulsed Low Dose Rate Radiation Therapy for Gastric Cancer Patients With Peritoneal Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yang Yang (Other)
Responsible Party: Sponsor-Investigator, Yang Yang, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLDR-RT-GC
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Radiotherapy; Radiotherapy Side Effect; Stomach Neoplasms
MeSH Terms: conditions — Radiation Injuries; Stomach Neoplasms | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Gastric cancer patients with peritoneal metastasis undergo pulsed low dose rate 3-dimensional conformal radiation therapy, QD, 5 days a week for 25 days. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: pulsed low dose rate radiation therapy

INTERVENTIONS:
Radiation: pulsed low dose rate radiation therapy — Pulsed low dose rate 3-dimensional conformal radiation therapy

SUMMARY:
This phase II trial studies the side effects and response of pulsed low dose rate radiation therapy in treating gastric cancer patients with peritoneal metastasis.

DETAILED DESCRIPTION:
This phase II trial studies the side effects and response of pulsed low dose rate radiation therapy in treating gastric cancer patients with peritoneal metastasis. Radiation therapy uses pulsed low dose rate high energy X rays to kill tumor cells and make less side effects than conventional 3-dimensional conformal radiation therapy. Palliative radiation therapy may help gastric cancer patients with peritoneal metastasis live more comfortably.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed gastric adenocarcinoma
* Patients must have metastasis tumor located within peritoneal cavity
* Tumor within the irradiated field is negatively impacting patient's quality of life or threatening catastrophic complication if left untreated as determined by the treating physician
* Patient is not a surgical candidate or tumor is not surgically resectable, as documented by surgical oncologist
* Patient is not a candidate for, or has not demonstrated a significant local response to chemotherapy, biologic, or other therapies
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 in the irradiated field
* Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to radiation simulation, postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential) and nonlactating, and men and women must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy completed
* Eastern Cooperative Oncology Group (ECOG) performance status determined to be between 0 and 3
* Absolute neutrophil count (ANC) >=1,000/ul
* Platelets (PLT) >=75,000/ul
* Subjects must sign a written informed consent and Health Insurance Probability and Accountability Act (HIPAA) consent prior to performance of study-specific procedures of assessments and must be willing to comply with treatment and follow-up

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy to the reirradiation target within 4 weeks prior to entering the study
* A history of ataxia telangiectasia or other documented history of radiation hypersensitivity
* Scleroderma or active connective tissue disease
* Active inflammatory bowel disease
* Serious, active infections requiring treatment with intravenous (IV) antibiotics
* Uncontrolled intercurrent illness including, but not limited to, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Side effects of pulsed low dose rate radiation therapy | Up to 30 days
  Number of participants with adverse events and the grade of adverse events. Graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Objective response | Up to 30 days
  Objective response of the target tumor were assessed using the Response Evaluation Criteria in Solid Tumor (RESICT) 1.1 criteria.
Palliative efficacy in terms of quality of life and pain levels | Up to 3 years
  Assessed using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 15 Palliative (QLQ-C15-PAL) and the Numeric Pain Scale. The mean and standard deviation will be estimated at each time point.
Duration of response | Up to 3 years
  Measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Assessed using the RESICT 1.1 criteria. Estimated using Kaplan-Meier curves.
Time to progression | Up to 3 years
  Assessed using the RECIST 1.1 criteria. Estimated using Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, MD,PhD,MSCR, Principal Investigator — The Comprehensive Cancer Center of Nanjing Drum Tower Hospital, Medical School of Nanjing University and Clinical Cancer Institute of Nanjing University
Locations (1):
- The Comprehensive Cancer Center of Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan J, Yang J, Yang Y, Ren W, Liu J, Gao S, Li S, Kong W, Zhu L, Yang M, Qian X, Liu B. Use of Pulsed Low-Dose Rate Radiotherapy in Refractory Malignancies. Transl Oncol. 2018 Feb;11(1):175-181. doi: 10.1016/j.tranon.2017.12.004. Epub 2018 Jan 4. PMID 29306203